CLINICAL TRIAL: NCT02717221
Title: An EGFR-TKIs Benefit Non-small Cell Lung Carcinoma Patients Identification Strategy and Treatment Response Using Molecular Imaging
Brief Title: In Vivo EGFR Molecular Classification and Treatment Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Xilin Sun, Chief, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14400
Record Dates: First submitted 2016-03-08; First posted 2016-03-23 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Molecular Imaging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 18F-MPG:EGFR+ (Experimental): Patients in this group had EGFR-activating mutant tumors and did not receive any treatment before this study.
  Interventions: Other: 18F-MPG
- 18F-MPG:post-TKI EGFR+ (Experimental): Patients with EGFR-activating mutant tumors were receiving EGFR-TKIs during this study.
  Interventions: Other: 18F-MPG
- 18F-MPG:post-chemo EGFR+ (Experimental): Patients with EGFR-activating mutant tumors were receiving chemotherapy during this study.
  Interventions: Other: 18F-MPG
- 18F-MPG:EGFR wild type (Experimental): Patients in this group had EGFR wild-type tumors and did not receive any treatment before this study.
  Interventions: Other: 18F-MPG
- 18F-MPG:post-chemo EGFR wild type (Experimental): Patients in this group had EGFR wild-type tumors and were receiving chemotherapy during this study.
  Interventions: Other: 18F-MPG
- 18F-MPG:unknown EGFR mutational status (Experimental): Patients without the EGFR mutational status measurement results and did not receive any treatments were classified in this group
  Interventions: Other: 18F-MPG

INTERVENTIONS:
Other: 18F-MPG — N-(3-chloro-4-fluorophenyl)-7-(2-(2-(2-(2-[18F] fluoroethoxy) ethoxy) ethoxy) ethoxy)-6-methoxyquinazolin-4-amine (18F-MPG)

SUMMARY:
The investigators developed 18F-MPG as a targeted molecular imaging agent for noninvasive and repeatable detecting EGFR-activating mutational status. And use 18F-MPG to monitor EGFR-TKIs and chemotherapy treatment efficiency.

DETAILED DESCRIPTION:
The goal of investigators were to evaluate the use of 18F-MPG as a novel PET/CT radiotracer to monitor EGFR-activating mutational status and identify EGFR-TKIs benefit NSCLC patients. the investigators want to evaluated the use of 18F-MPG in lung cancer imaging in adult NSCLC patients with different EGFR mutational status of primary and metastatic cancers. And the investigators want to evaluated the use of 18F-MPG in adult NSCLC patients with EGFR mutational status received non-treatment, EGFR-TKIs and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC
* 18 years or older
* A life expectancy of at least 12 weeks
* Presence of a malignant lesion within the chest of at least 0.5 cm diameter as measured by computed tomography (CT)
* Written informed consent

Exclusion Criteria:

* Claustrophobia
* Pregnancy
* Metal implants in the thorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-11; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
tumor SUVmax value of 18F-MPG PET/CT Imaging | at time of imaging
  To quantify the accumulation, a volume of interest using a 3-D sphere, was placed over the primary lung tumor, lymph nodes and distant metastases avoiding necrosis, blood vessels and normal lung tissue as much as possible on a workstation (Advantage Workstation 4.6; GE Healthcare). The maximum standard uptake value (SUVmax) normalized to body weight (kBq/mL) was calculated within the region of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Baozhong Shen, M.D., Study Chair — The Fourth Hospital of Harbin Medical University
Locations (1):
- TOF-PET/CT/MR center of the Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Slobbe P, Windhorst AD, Stigter-van Walsum M, Smit EF, Niessen HG, Solca F, Stehle G, van Dongen GA, Poot AJ. A comparative PET imaging study with the reversible and irreversible EGFR tyrosine kinase inhibitors [(11)C]erlotinib and [(18)F]afatinib in lung cancer-bearing mice. EJNMMI Res. 2015 Mar 20;5:14. doi: 10.1186/s13550-015-0088-0. eCollection 2015. PMID 25853020
- [Background] Abourbeh G, Itamar B, Salnikov O, Beltsov S, Mishani E. Identifying erlotinib-sensitive non-small cell lung carcinoma tumors in mice using [(11)C]erlotinib PET. EJNMMI Res. 2015 Feb 12;5:4. doi: 10.1186/s13550-014-0080-0. eCollection 2015. PMID 25853010
- [Background] Petrulli JR, Sullivan JM, Zheng MQ, Bennett DC, Charest J, Huang Y, Morris ED, Contessa JN. Quantitative analysis of [11C]-erlotinib PET demonstrates specific binding for activating mutations of the EGFR kinase domain. Neoplasia. 2013 Dec;15(12):1347-53. doi: 10.1593/neo.131666. PMID 24403856
- [Background] Yeh SH, Lin CF, Kong FL, Wang HE, Hsieh YJ, Gelovani JG, Liu RS. Molecular imaging of nonsmall cell lung carcinomas expressing active mutant EGFR kinase using PET with [(124)i]-morpholino-IPQA. Biomed Res Int. 2013;2013:549359. doi: 10.1155/2013/549359. Epub 2013 Jul 17. PMID 23956990
- [Background] Yeh HH, Ogawa K, Balatoni J, Mukhapadhyay U, Pal A, Gonzalez-Lepera C, Shavrin A, Soghomonyan S, Flores L 2nd, Young D, Volgin AY, Najjar AM, Krasnykh V, Tong W, Alauddin MM, Gelovani JG. Molecular imaging of active mutant L858R EGF receptor (EGFR) kinase-expressing nonsmall cell lung carcinomas using PET/CT. Proc Natl Acad Sci U S A. 2011 Jan 25;108(4):1603-8. doi: 10.1073/pnas.1010744108. Epub 2011 Jan 10. PMID 21220318
- [Background] Pal A, Balatoni JA, Mukhopadhyay U, Ogawa K, Gonzalez-Lepera C, Shavrin A, Volgin A, Tong W, Alauddin MM, Gelovani JG. Radiosynthesis and initial in vitro evaluation of [18F]F-PEG6-IPQA--a novel PET radiotracer for imaging EGFR expression-activity in lung carcinomas. Mol Imaging Biol. 2011 Oct;13(5):853-61. doi: 10.1007/s11307-010-0408-8. PMID 20859697
- [Background] Zannetti A, Iommelli F, Speranza A, Salvatore M, Del Vecchio S. 3'-deoxy-3'-18F-fluorothymidine PET/CT to guide therapy with epidermal growth factor receptor antagonists and Bcl-xL inhibitors in non-small cell lung cancer. J Nucl Med. 2012 Mar;53(3):443-50. doi: 10.2967/jnumed.111.096503. Epub 2012 Feb 13. PMID 22331221
- [Background] Gerbaudo VH, Kim CK. PET Imaging-Based Phenotyping as a Predictive Biomarker of Response to Tyrosine Kinase Inhibitor Therapy in Non-small Cell Lung Cancer: Are We There Yet? Nucl Med Mol Imaging. 2017 Mar;51(1):3-10. doi: 10.1007/s13139-016-0453-6. Epub 2016 Oct 11. PMID 28250852
- [Background] Nakamura Y, Ohler ZW, Householder D, Nagaya T, Sato K, Okuyama S, Ogata F, Daar D, Hoa T, Choyke PL, Kobayashi H. Near Infrared Photoimmunotherapy in a Transgenic Mouse Model of Spontaneous Epidermal Growth Factor Receptor (EGFR)-expressing Lung Cancer. Mol Cancer Ther. 2017 Feb;16(2):408-414. doi: 10.1158/1535-7163.MCT-16-0663. Epub 2016 Nov 15. PMID 28151706